CLINICAL TRIAL: NCT00097721
Title: A Phase II Open Label Study of E7389 (Halichondrin B Analog) in Patients With Advanced/Metastatic Breast Cancer Previously Treated With Chemotherapy Including An Anthracycline and A Taxane
Brief Title: A Study of E7389 in Advanced/Metastatic Breast Cancer Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E7389-A001-201
Record Dates: First submitted 2004-11-29; First posted 2004-11-30 (Estimated); Results first posted 2013-03-15 (Estimated); Last update posted 2013-04-22 (Estimated); Status verified 2013-04

CONDITIONS: Breast Neoplasms
Keywords: breast neoplasm; breast cancer; breast tumor
MeSH Terms: conditions — Breast Neoplasms | interventions — eribulin

ARMS (1):
- E7389 (Experimental)
  Interventions: Drug: E7389

INTERVENTIONS:
Drug: E7389 — The first cohort of subjects were to receive E7389 1.4 mg/m^2 as an intravenous (IV) bolus on Days 1, 8, and 15 of a 28-day cycle. A second cohort of subjects was added and were to receive E7389 1.4 mg/m^2 as an IV bolus on Days 1 and 8 of a 21-day cycle.

SUMMARY:
The purpose of this study is to determine if E7389 is a safe and effective treatment for advanced/metastatic breast cancer.

DETAILED DESCRIPTION:
The primary objective is to determine the response rate (RR) to E7389 monotherapy administered as an IV bolus of 1.4 mg/m^2 on Days 1, 8, and 15 of a 28-Day cycle and on Days 1 and 8 of a 21-day cycle in patients with advanced/metastatic breast cancer treated with chemotherapy including an anthracycline and a taxane, with previously documented progression during or within six months following the last dose of prior chemotherapy.

The secondary objectives are to evaluate:

* The safety and tolerability of E7389 monotherapy in this patient population;
* The antitumor activity of E7389 as determined by duration of response, time to progression, and overall survival;
* Quality of life measured by the Functional Assessment of Cancer Therapy-Breast (FACT-B) questionnaire/tumor-related symptom improvement or worsening measured by pain intensity on a visual analog scale (VAS), analgesics consumption, weight changes and performance status (PS);
* Tumor pharmacogenetics and their possible relationship to response (assessment of beta-tubulin isotype mRNA on biopsy sample) in patients who have signed a separate consent form

ELIGIBILITY:
Inclusion Criteria:

* Female patients with histologically or cytologically confirmed carcinoma of the breast
* Patients with advanced/metastatic disease that is not amenable to curative therapy (either surgery or radiation therapy)
* Patients must have measurable disease by the RECIST criteria, defined as at least one lesion that can be accurately measured in at least one diameter (at least 10 mm in longest diameter (LD) by spiral computer tomography (CT) scan, or at least 20 mm by standard techniques; If the only measurable lesion is a lymph node, it must measure at least 20 mm in LD. If a single lesion is identified as the target lesion, a cytological or histological confirmation of breast carcinoma is required.
* Patients must have had prior treatment with an anthracycline and a taxane (either sequential or in combination) and may have had prior treatment with other agents as well.
* Patients must have progressed within six months of the last dose of chemotherapy, or experienced disease progression while receiving chemotherapy for advanced/metastatic disease.
* Resolution of all chemotherapy or radiation-related toxicities to less than grade 1 severity
* Age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) Performance Status (APPENDIX 4) of 0 or 1
* Life expectancy of ≥ 3 months
* Adequate renal function as evidenced by serum creatinine ≤ 1.5 mg/dL or calculated creatinine clearance ≥ 50 mL/minute (min) per the Cockcroft and Gault formula
* Adequate bone marrow function as evidenced by absolute neutrophil count (ANC) ≥ 1.5 x 10^9/L, hemoglobin ≥ 10.0 g/dL (a hemoglobin <10.0 g/dL would be acceptable if it can be corrected by growth factor or transfusion), and platelet count ≥ 100 x 10^9/L
* Adequate liver function as evidenced by bilirubin ≤ 1.5 mg/dL and alkaline phosphatase, alanine transaminase (ALT), and aspartate transaminase (AST) ≤ 3 times the upper limits of normal (ULN) (in the case of liver metastases ≤ 5 x ULN)
* Patients willing and able to complete the FACT-B questionnaire, Analgesic Diary, Pain VAS, and the tumor-related symptomatic assessment
* Patients willing and able to comply with the study protocol for the duration of the study
* A sample from the diagnostic biopsy (paraffin block) must be available
* Written informed consent prior to any study-specific screening procedures with the understanding that the patient may withdraw consent at any time without prejudice

Exclusion Criteria:

* Patients who have received chemotherapy, radiation, hormonal therapy, or Herceptin within 2 weeks of E7389 treatment start
* Radiation therapy encompassing > 10% of marrow
* Failure to recover from any chemotherapy related or other therapy related toxicity at study entry that is deemed to be clinically significant by the study investigator
* Prior treatment with Mitomycin C or nitrosoureas
* Prior high dose chemotherapy with hematopoietic stem cell rescue in the past two years
* Pulmonary lymphangitic involvement that results in pulmonary dysfunction requiring active treatment, including the use of oxygen
* Active symptomatic brain metastasis; Patients with central Nervous System (CNS) metastasis are considered eligible if they have completed local therapy and discontinued from corticosteroids for at least two weeks before starting treatment with E7389
* Patients with meningeal carcinomatosis
* Patients who require therapeutic anti-coagulant therapy with Warfarin or related compounds; Mini dose warfarin for catheter related thrombosis prophylaxis is permitted
* Women who are pregnant or breast-feeding; Women of childbearing potential with either a positive pregnancy test at Screening or no pregnancy test. Women of childbearing potential unless (1) surgically sterile or (2) using adequate measures of contraception in the opinion of the Investigator. Postmenopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential.
* Severe /uncontrolled intercurrent illness/infection
* Significant cardiovascular impairment (history of congestive heart failure > NYHA grade II, unstable angina or myocardial infarction within the past six months, or serious cardiac arrhythmia)
* Patients with organ allografts
* Patients with known positive HIV status
* Patients who have had a prior malignancy, other than carcinoma in situ of the cervix, or non-melanoma skin cancer, unless the prior malignancy was diagnosed and definitively treated ≥ 5 years previously with no subsequent evidence of recurrence
* Patients with pre-existing neuropathy > Grade 1
* Patients with a hypersensitivity to halichondrin B and/or halichondrin B chemical derivative
* Patients who participated in a prior E7389 clinical trial
* Patients with other significant disease or disorders that, in the Investigator's opinion, would exclude the patient from the study

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2004-09; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dale Shuster, Ph.D., Study Director — Eisai Inc.
Locations (16):
- United States (16):
  - Jonesboro, Arkansas
  - Deer Park, California
  - La Verne, California
  - Pasadena, California
  - Pomona, California
  - Brooksville, Florida
  - New Port Richey, Florida
  - Plantation, Florida
  - New Orleans, Louisiana
  - Southaven, Mississippi
  - Missoula, Montana
  - Syracuse, New York
  - Middletown, Ohio
  - Memphis, Tennessee
  - Amarillo, Texas
  - Richardson, Texas

REFERENCES:
- [Derived] Muss H, Cortes J, Vahdat LT, Cardoso F, Twelves C, Wanders J, Dutcus CE, Yang J, Seegobin S, O'Shaughnessy J. Eribulin monotherapy in patients aged 70 years and older with metastatic breast cancer. Oncologist. 2014 Apr;19(4):318-27. doi: 10.1634/theoncologist.2013-0282. Epub 2014 Mar 28. PMID 24682463
- See also: Official company website — http://www.eisai.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was recruited at 23 centers in U.S. during the period of Nov 2004 to Nov 2006.
Groups:
- E7389 28 Day Schedule: E7389 1.4 mg/m^2 intravenous bolus on Days 1, 8 and 15 of a 28 day cycle.
- E7389 21 Day Schedule: E7389 1.4 mg/m^2 intravenous bolus on Days 1 and 8 of a 21 day cycle.
Period: Overall Study
Arm/Group | E7389 28 Day Schedule | E7389 21 Day Schedule
Started | 71 (The number started is all enrolled subjects.BL Characteristics consists of Safety Population.) | 33
Completed | 0 | 0
Not Completed | 71 | 33
Not completed — Adverse Event | 8 | 1
Not completed — Withdrawal by Subject | 6 | 1
Not completed — Progressive Disease | 55 | 27
Not completed — Physician Decision | 1 | 3
Not completed — Reason not given | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | E7389 28 Day Schedule | E7389 21 Day Schedule | Total
Number analyzed (Participants) | 70 | 33 | 103
Age Continuous [Mean (Standard Deviation); unit: years] | 55.9 (10.7) | 54.5 (10.99) | 55.4 (10.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 70 | 33 | 103
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 6 | 11
  White | 51 | 21 | 72
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
  Hispanic/Latino | 9 | 3 | 12
  Other | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate Based on Response Evaluation Criteria in Solid Tumors (RECIST)
Description: Defined as the percentage of subjects with CR or PR from the start of treatment until disease progression or recurrence. Lesions measured by computed tomography (CT) scan and magnetic resonance imaging (MRI). Objective response rate: complete response (CR-disappearance of all lesions)+ partial response (PR-30% decrease in lesion diameter), Progressive Disease (PD-20% increase in lesion diameter), stable disease (SD-neither shrinkage nor increase of lesions).
Time Frame: Confirmed 4 to 8 weeks after first observed
Population: Per Protocol Population (Independent Reviewer Assessment)
Measure: Number; unit: percentage of participants
Arm/Group | E7389 28 Day Schedule | E7389 21 Day Schedule
Number analyzed (Participants) | 59 | 28
percentage of participants
  Complete Response: | 0 | 0
  Partial Response | 10.2 | 14.3

2. Secondary Outcome: Duration of Response
Description: Measured from the time measurement criteria were met for complete response (CR) or partial response (PR) (whichever was first recorded) until the first date that recurrent progressive disease was objectively documented (taking as a reference for progressive disease the smallest measurements recorded since the treatment started).
Time Frame: From CR or partial response PR (whichever recorded first) to date of recurrent or progressive disease
Population: Intent to Treat/Safety Population (Investigator Assessment)
Measure: Median (Full Range); unit: days
Arm/Group | E7389 28 Day Schedule | E7389 21 Day Schedule
Number analyzed (Participants) | 70 | 33
days | 204 [93 to 428] | 121 [83 to 277]

3. Secondary Outcome: Progression Free Survival
Description: Defined as the time from start of study drug administration until progressive disease or death from any cause during the study period in the absence of disease progression.
Time Frame: From start of study drug administration to progressive disease or death
Population: Per Protocol Population (Investigator Assessment)
Measure: Median (Full Range); unit: days
Arm/Group | E7389 28 Day Schedule | E7389 21 Day Schedule
Number analyzed (Participants) | 59 | 28
days | 57 [1 to 413] | 86 [1 to 453]

4. Secondary Outcome: Overall Survival
Description: Defined as the time from the start of study drug administration until death from any cause
Time Frame: From start of study drug administration to death
Population: Per Protocol Population (Investigator Assessment)
Measure: Median (Full Range); unit: days
Arm/Group | E7389 28 Day Schedule | E7389 21 Day Schedule
Number analyzed (Participants) | 59 | 28
days | 239 [15 to 826] | NA [18 to 620] — This data point is not available due to insufficient number of deaths.

5. Secondary Outcome: Change From Baseline to Study Termination in Quality of Life Measures Using Functional Assessment of Cancer Therapy-Breast (FACT-B) Scores
Description: The FACT-B questionnaire consists of 36 questions each scored from 0-4. The total score is calculated by summing these scores. The total possible range is from 0 to 144. The higher scores indicate a better health-related quality of life. This measures emotional, functional, physical, and social well being as well as concerns specific to patients with breast cancer.
Time Frame: At Screening, Day 1 of each cycle, and 30 days after last dose of study drug
Measure: Median (Full Range); unit: units on a scale
Arm/Group | E7389 28 Day Schedule | E7389 21 Day Schedule
Number analyzed (Participants) | 40 | 21
units on a scale
  Change From Baseline | -2.2 [-30 to 34] | 0 [-34 to 37.8]
  Baseline Score | 102.0 [56.0 to 140.6] | 101.0 [57.9 to 138.0]
  Study Termination Score | 104.3 [50.0 to 143.0] | 98.4 [65.0 to 139.0]

ADVERSE EVENTS:
Arm/Group | E7389 28 Day Schedule | E7389 21 Day Schedule
Serious Adverse Events (participants affected / at risk) | 23/70 | 18/33
Other Adverse Events (participants affected / at risk) | 69/70 | 33/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | E7389 28 Day Schedule (N=70) | E7389 21 Day Schedule (N=33)
Febrile Neutropenia (Blood and lymphatic system disorders) | 2 | 1
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Inner Ear Disorder (Ear and labyrinth disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 1 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 1 | 0
Ascites (Gastrointestinal disorders) | 1 | 0
Diarrhea (Gastrointestinal disorders) | 1 | 0
Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 0 | 1
Disease Progression (General disorders) | 3 | 1
Mucosal Inflammation (General disorders) | 1 | 0
Pain (General disorders) | 0 | 3
Pyrexia (General disorders) | 3 | 2
Hepatic Failure (Hepatobiliary disorders) | 0 | 1
Bacterial Pyelonephritis (Infections and infestations) | 1 | 1
Bronchiectasis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Catheter Related Infection (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 1
Meningitis Listeria (Infections and infestations) | 1 | 0
Neutropenic Sepsis (Infections and infestations) | 1 | 0
Oropharyngeal Candidiasis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Upper Respiratory Tract (Infections and infestations) | 1 | 0
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 5 | 1
Failure to Thrive (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Groin Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Malignant Neoplasm Progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Confusional State (Psychiatric disorders) | 1 | 0
Hydronephrosis (Renal and urinary disorders) | 1 | 0 (0)
Female Genital Tract Fistula (Reproductive system and breast disorders) | 0 | 1
Chronic Obstructive Pulmonary (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0
Swelling Face (Skin and subcutaneous tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | E7389 28 Day Schedule (N=70) | E7389 21 Day Schedule (N=33)
Anemia (Blood and lymphatic system disorders) | 34 | 7
Leukocytosis (Blood and lymphatic system disorders) | 4 | 0
Leukopenia (Blood and lymphatic system disorders) | 22 | 6
Neutropenia (Blood and lymphatic system disorders) | 54 | 24
Thrombocytopenia (Blood and lymphatic system disorders) | 8 | 1
Tachycardia (Cardiac disorders) | 9 | 1
Lacrimation Increased (Eye disorders) | 4 | 2
Vision Blurred (Eye disorders) | 5 | 1
Abdominal Discomfort (Gastrointestinal disorders) | 6 | 0
Abdominal Distention (Gastrointestinal disorders) | 5 | 3
Abdominal Pain (Gastrointestinal disorders) | 9 | 5
Abdominal Pain Upper (Gastrointestinal disorders) | 4 | 1
Constipation (Gastrointestinal disorders) | 25 | 10
Diarrhea (Gastrointestinal disorders) | 11 | 8
Dry Mouth (Gastrointestinal disorders) | 5 | 4
Dyspepsia (Gastrointestinal disorders) | 8 | 4
Nausea (Gastrointestinal disorders) | 32 | 14
Oral Pain (Gastrointestinal disorders) | 4 | 1
Stomach Discomfort (Gastrointestinal disorders) | 0 | 2
Stomatitis (Gastrointestinal disorders) | 13 | 6
Vomiting (Gastrointestinal disorders) | 13 | 8
Asthenia (General disorders) | 3 | 3
Chest Discomfort (General disorders) | 5 | 1
Chest Pain (General disorders) | 3 | 4
Chills (General disorders) | 3 | 3
Fatigue (General disorders) | 41 | 19
Mucosal Inflammation (General disorders) | 5 | 1
Edema (General disorders) | 4 | 1
Edema Peripheral (General disorders) | 17 | 5
Pain (General disorders) | 8 | 5
Pyrexia (General disorders) | 23 | 8
Infection (Infections and infestations) | 1 | 2
Sinusitis (Infections and infestations) | 0 | 2
Upper Respiratory Tract Infection (Infections and infestations) | 3 | 7
Urinary Tract Infection (Infections and infestations) | 9 | 5
Aspartate Aminotransferase Increased (Investigations) | 0 | 3
Blood Alkaline Phosphatase Increased (Investigations) | 1 | 3
Breath Sounds Abnormal (Investigations) | 2 | 2
White Blood Cell Count Decreased (Investigations) | 1 | 2
Alanine Aminotransferase Increased (Investigations) | 0 | 2
Anorexia (Metabolism and nutrition disorders) | 17 | 6
Decreased Appetite (Metabolism and nutrition disorders) | 5 | 4
Dehydration (Metabolism and nutrition disorders) | 11 | 3
Hypoalbuminemia (Metabolism and nutrition disorders) | 4 | 1
Hypokalemia (Metabolism and nutrition disorders) | 12 | 7
Hypomagnesemia (Metabolism and nutrition disorders) | 6 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 9 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 9 | 5
Bone Pain (Musculoskeletal and connective tissue disorders) | 9 | 3
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 6 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 3
Pain Extemity (Musculoskeletal and connective tissue disorders) | 10 | 0
Shoulder Pain (Musculoskeletal and connective tissue disorders) | 4 | 2
Coordination Abnormal (Nervous system disorders) | 4 | 0
Dizziness (Nervous system disorders) | 10 | 7
Dysgeusia (Nervous system disorders) | 7 | 3
Headache (Nervous system disorders) | 12 | 11
Hypoaesthesia (Nervous system disorders) | 2 | 3
Neuropathy (Nervous system disorders) | 5 | 2
Neuropathy Peripheral (Nervous system disorders) | 14 | 7
Paraesthesia (Nervous system disorders) | 5 | 2
Peripheral Sensory Neuropathy (Nervous system disorders) | 6 | 1
Tremor (Nervous system disorders) | 2 | 2
Insomnia (Psychiatric disorders) | 6 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 7
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 19 | 8
Dyspnea Exertional (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Pharyngolarygeal Pain (Respiratory, thoracic and mediastinal disorders) | 6 | 6
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 4 | 2
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dysuria (Renal and urinary disorders) | 4 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 31 | 14
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritis (Skin and subcutaneous tissue disorders) | 3 | 4
Skin Lesion (Skin and subcutaneous tissue disorders) | 1 | 2
Hot Flush (Vascular disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No